CLINICAL TRIAL: NCT02112149
Title: Effect of the LIVESTRONG at the YMCA Exercise Program on Cancer Related Outcomes in Cancer Survivors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1301011291
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Body Composition; Exercise; Survivorship
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LIVESTRONG Program (Experimental): Participants randomized to the LIVESTRONG exercise program will attend a 12-week LIVESTRONG Program at one of the participating YMCA's in the greater Boston area or CT. We will have monthly teleconferences to discuss the study, recruitment, and the exercise program. Lastly, throughout the 12-week program, participants will record their attendance at the LIVESTRONG program as well as any exercise done outside of the program. We will provide them with a Physical Activity Log book to record their exercise.
  Interventions: Behavioral: LIVESTRONG
- Wait-List Control (No Intervention): Baseline data will be collected from all study participants before randomization. If a participant is randomized to wait-list control, then he/she will be told that he/she will start the LIVESTRONG program after three months and after he/she returns to Yale or DFCI to complete the 3-month clinic visit.

INTERVENTIONS:
Behavioral: LIVESTRONG — The LIVESTRONG at the YMCA is a twelve-week, small group (< 16 participants) program designed for adult cancer survivors. YMCA fitness instructors work with each participant to fit the program to their individual needs. The instructors are trained in the elements of cancer, post rehabilitation exercise and supportive cancer care. There are two YMCA fitness instructors overseeing each exercise session. Each session is 90 min in duration, twice per week, for 12-wks (total of 24 sessions). Each session begins with a warm-up, then aerobic exercise (e.g., treadmill) and resistance training exercises, followed by a cool-down period, and follows the recommendations of the American College of Sports Medicine.
  Arms: LIVESTRONG Program

SUMMARY:
The proposed study is a randomized trial evaluating the impact of the 12-week LIVESTRONG exercise program vs. waitlist control on cancer-related outcomes in 200 cancer survivors.

DETAILED DESCRIPTION:
The proposed study is a randomized trial evaluating the impact of the 12-week LIVESTRONG exercise program vs. waitlist control on cancer-related outcomes in 200 cancer survivors. Participants will undergo baseline testing at Dana-Farber or Yale, including administration of questionnaires to assess quality of life and the presence of cancer and treatment-related symptoms, fasting blood draw, and evaluation of body composition (using dual energy X-ray absorptiometry (DEXA). Participants will then take part in the 12-week LIVESTRONG Program or will be assigned to a wait-list control group. All measurements will be repeated at Dana-Farber or Yale after the 12-week exercise program or control period.

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis excluding non-melanoma skin cancer
* Physically able to exercise
* Able to complete forms and understand instructions in English
* Agrees to be randomly assigned to either exercise or wait-list control group
* Willing and able to attend one of the LIVESTRONG at the YMCA programs for 12 weeks
* Willing and able to complete the baseline and 3-month clinic visits

Exclusion Criteria:

* > 80 years of age
* < 18 years of age
* Recent (past 6 months) stroke/myocardial infarction or congestive heart failure/documented ejection fraction < 40%
* Plans to undergo a major surgical procedure in the next 6 months
* Presence of dementia or major psychiatric disease that would preclude participation in a group-based exercise program
* Pregnant women or women intending to become pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity Level | 3 months
  Modifiable Physical Activity Questionnaire will be used to assess physical activity levels at baseline and 3-months to examine whether the LIVESTRONG program led to maintenance or further increases in physical activity levels compared with participants randomized to control.

SECONDARY OUTCOMES:
Change in Body Fat Percentage | 3 months
  Dual-energy X-ray absorptiometry (DEXA) scans will be used to assess body fat percentage, lean body mass, and bone mineral density at baseline and 3-months. Study participants will receive a copy of their 3-month DEXA report.
Change in Lean Body Mass | 3 months
  Dual-energy X-ray absorptiometry (DEXA) scans will be used to assess body fat percentage, lean body mass, and bone mineral density at baseline and 3-months. Study participants will receive a copy of their 3-month DEXA report.
Change in Bone Mineral Density | 3 months
  Dual-energy X-ray absorptiometry (DEXA) scans will be used to assess body fat percentage, lean body mass, and bone mineral density at baseline and 3-months. Study participants will receive a copy of their 3-month DEXA report.
Change in Body Mass Index (BMI) | 3 months
  Height and weight will be measured at baseline and 3-months. Participants will be weighed in light indoor clothing, without shoes, rounding up to the nearest 0.1 kg; height will be measured without shoes, using a stadiometer, rounding up to the nearest 0.1 cm. BMI will be calculated using the formula: kg/m2. All measures will be performed and recorded twice in succession.
Change in Blood Biomarkers | 12 weeks
  Fasting blood (> 12 hours) will be collected at baseline and 12 weeks for measurement of insulin, c-reactive protein, leptin and adiponectin, which are biomarkers that have been linked to cancer prognosis in prior studies.

OTHER OUTCOMES:
Change in Walk Distance | 12 weeks
  All participants will undergo a 6MWT at baseline and after the 12-week protocol period. Participants will wear tennis shoes and will walk indoors along a long, flat, straight, enclosed corridor, on a flat surface for 6 minutes. They will be instructed to walk continuously along an area at least 50 feet in length, back and forth, for 6 minutes.
Change in Quality of Life | 12 weeks
  Quality of Life (QOL) will be measured using the Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire (version 3) as well as the PROMISE Q. Breast cancer survivors will also complete the FACT-B-ES form that assesses endocrine-related symptoms specific to breast cancer. Additionally, fatigue will be assessed through the FACT-Fatigue Scale, which consists of 13 items designed to assess fatigue in terms of its intensity and interference with performing everyday functions.
Lymphedema Questionnaire | 12 weeks
  Breast cancer survivors will complete a validated Norman Lymphedema Questionnaire. Previous methodologically strong studies have shown exercise, including upper body resistance/strength training, to decrease the risk of exacerbation of lymphedema as well as severity of lymphedema symptoms in breast cancer survivors randomized to a twice-weekly year long strength training program compared with breast cancer survivors randomized to control. Given these findings, breast cancer survivors with lymphedema will not be excluded from participation in the study. However, MD consent to exercise will be obtained from her oncologist.
Change in Breast Cancer Prevention Trial Symptom Checklist | 3 months
  The Breast Cancer Prevention Trial Symptom Checklist Short Form is a symptom checklist that will be completed by all study participants at baseline and 3-months to assess side effects/symptoms related to cancer surgery and treatment and how exercise may improve or prevent some of these symptoms. Symptoms such as lymphedema, neuropathy, and arthralgias will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda L Irwin, PhD, MPH, Principal Investigator — Yale University; Jennifer A Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Dana-Farber Cancer Institute, Boston, Massachusetts